CLINICAL TRIAL: NCT03451669
Title: Thermal Camera Detection of Ventriculoperitoneal Shunt Flow
Acronym: Infrared Shunt
Status: Completed | Type: Observational
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Other Study IDs: 827169
Record Dates: First submitted 2018-02-23; First posted 2018-03-02 (Actual); Last update posted 2020-05-11 (Actual); Status verified 2020-05

CONDITIONS: Hydrocephalus
MeSH Terms: conditions — Hydrocephalus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Shunt suspected to be functioning
- Shunt suspected to not be functioning

SUMMARY:
There have been reports in the past of using thermal cameras to demonstrate flow in the tubing as a surrogate of proper shunt function. This was shown to have almost 90% accuracy at determining proper functioning but required expensive equipment that was not universally available. There is now smart phone based thermal camera technology (Flir One: http://www.flir.com/flirone/) that could make this technique widely available for health care use. The goal of the study is to determine if this device can demonstrate flow in the distal tubing of a VP shunt.

ELIGIBILITY:
Inclusion Criteria:

* Patients with known VP shunt
* Status of shunt function known.
* Patients with well healed wounds (no immediately post op patients)

Exclusion Criteria:

* Patients in urgent need of shunt revision
* Age less than 18

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Adult patients with VP shunts at the University of Pennsylvania, Department of Neurosurgery
Sampling Method: Non-Probability Sample
Enrollment: 2 (Actual)
Dates: Start 2018-04-16 (Actual); Primary Completion 2019-11-30 (Actual); Study Completion 2019-12-02 (Actual)

PRIMARY OUTCOMES:
Determine if a smartphone based thermal camera can determine flow in the distal tubing of a VP shunt. | 3 years

CONTACTS AND LOCATIONS:
Locations (1):
- University of Pennsylvania Medical Center, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No